CLINICAL TRIAL: NCT06070857
Title: A Randomized, Double-blind, Placebo-Controlled, Single-Centre,Single Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of LV232 Capsules in Chinese Healthy Volunteers
Brief Title: Study of the Safety, Tolerability, and Pharmacokinetics of LV232 Capsules in Chinese Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LV232-01
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects
Keywords: LV232; Phase I; dose-escalation; Tolerability; Pharmacokinetic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LV232 (Experimental): Subjects will receive LV232 orally for single dose.
  Interventions: Drug: LV232
- Placebo (Experimental): Subjects will receive placebo orally for single dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LV232 — Drug: LV232 1mg,2mg,4mg,8mg,15mg,25mg,40mg,60mg,90mg and 120mg
  Arms: LV232
Drug: Placebo — Placebo:1mg,2mg,4mg,8mg,15mg,25mg,40mg,60mg,90mg and 120mg
  Arms: Placebo

SUMMARY:
The study consists of 10 dose groups, 8 subjects in each group (male or female), randomly assigned to study drug or placebo group to evaluate the safety, tolerability and pharmacokinetics characteristics.

DETAILED DESCRIPTION:
The dose levels are planned at 1 mg, 2 mg, 4 mg, 8 mg, 15 mg, 25 mg,40 mg, 60 mg ,90 mg and 120mg. 6 subjects in each group will receive LV232 tablets and 2 subjects will receive placebo. The subject number of single dose group may increase or decrease depending on the safety and PK data obtained.1 mg dose group will be given by sentinel administration (i.e. 1 study drug, 1 placebo). Subjects who receive sentinel administration will be observed for 48 hours and investigator will evaluate the safety parameters (including symptoms, vital signs, physical examination, etc.).Based on observed tolerability and safety data or obtained PK data, adjustments are allowed at all dose levels in the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 45 years old, males or females;
2. Body weight no less than 50.0 kg for male, no less than 45.0 kg for female,Body Mass Index of 19.0 to 26.0kg/m2;
3. Physical examination, vital signs examination, laboratory examination, electrocardiogram examination and B-ultrasound examination results were normal or abnormal without clinical significant;
4. Subjects who are willing to take effective contraceptive during the study and within 3 months after the study completed;
5. Subjects who are able to understand and follow study plans and instructions; Subjects who have voluntarily decided to participate in this study, and signed the informed consent form.

Exclusion Criteria:

1. Subjects with hypersensitivity to LV232 or any of the excipients;
2. Subjects with allergic diseases or allergic constitution;
3. Subjects with skin diseases or a history of skin allergies;
4. Subjects with central nervous system, cardiovascular system, gastrointestinal, respiratory system, urinary, Hematologic System, metabolic disorders that require medical intervention or other diseases (such as psychiatric history) that are not suitable for clinical trials;
5. Blood donation or blood loss ≥ 400 mL within 3 months , or have a history of blood product use history
6. Subjects who have participated in clinical trials of other drugs within 3 months before screening;
7. Subjects who have taken any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or health products orally within 2 weeks before screening;
8. Drug or alcohol addicts within 1 year prior to screening, who drink at least twice a day or more than 14 units per week, or who are addicted to alcohol (1 unit ≈200 mL beer with 5% alcohol content, 25 mL spirits with 40% alcohol content or 85 mL wine with 12% alcohol content);
9. Subjects who smoked more than 10 cigarettes or equivalent amounts of tobacco a day within one year before screening;
10. Subjects who can't quit smoking and drinking during the experiment;
11. Subjects who are positive for hepatitis B virus surface antigen, hepatitis C virus antibody, Treponema pallidum antibody (TPPA) or human immunodeficiency virus antibody (Anti-HIV);
12. Abnormal and clinically significant chest radiographs (anteroposterior);
13. B ultrasound examination showed moderate to severe fatty liver;
14. Pregnant or lactating woman or male subjects whose spouse has a child care plan within 3 months;
15. The investigator believes that there are other factors that are not suitable for participating in this trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 7 days after treatment
  Incidence of Treatment-Emergent Adverse Events
Cmax | 48 hours after administration
  maximum observed plasma concentration
AUC0-t | 48 hours after administration
  area under the plasma concentration time curve from time zero to the last
AUC0-∞ | 48 hours after administration
  area under the plasma concentration time curve from time zero to infinity
AUC0-24h | 48 hours after administration
  area under the plasma concentration time curve from time zero to 24 hours
Tmax | 48 hours after administration
  time at which Cmax occurs
t1/2 | 48 hours after administration
  half life of elimination
CL/F | 48 hours after administration
  apparent clearance
Vd/F | 48 hours after administration
  apparent volume of distribution during the terminal phase
Ke | 48 hours after administration
  elimination rate constant
MRT | 48 hours after administration
  mean Resident Time
BP | 48 hours after administration
  Blood Plasma Ratio
BRPP | 48 hours after administration
  binding rate of plasma protein

SECONDARY OUTCOMES:
structural of metabolites | From time zero up to 96 hours post-dose following oral administration
  Structure of main metabolites of LV232 in plasma, feces and urine
Ae | From time zero up to 96 hours post-dose following oral administration
  Cumulative excretion of LV232 and major metabolites in feces and urine
Fe% | From time zero up to 96 hours post-dose following oral administration
  Percentage of LV232 and major metabolites in feces and urine
CLr | From time zero up to 72 hours post-dose following oral administration
  renal clearance rate
Genetic polymorphisms in drug metabolism | Before administration
  Influence of genetic polymorphisms in drug metabolism enzymes on pharmacokinetics and safety

CONTACTS AND LOCATIONS:
Overall Officials: Chen Yu, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No